CLINICAL TRIAL: NCT00597974
Title: Evaluation of Neurological Outcome in Patients Undergoing Cerebral Angiography and Revascularization Using Angioplasty and Stent-Supported Angioplasty
Brief Title: Neurological Outcome With Carotid Artery Stenting
Acronym: CAS
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eric J. Heyer, MD, PhD, Professor of Clinical Anesthesiology, Columbia University
Other Study IDs: AAAA2389
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Carotid Artery Disease; Carotid Artery Stenosis; Stroke; Transient Ischemic Attack
Keywords: carotid artery stenosis; Neuropsychological tests; Stroke; Transient ischemia; Stenting
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Ischemic Attack, Transient | interventions — Angioplasty; Stents; Cerebral Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma serum DNA (obtained via buccal samples using a buccal cell collection swab)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients having angioplasty (case): Patients undergoing carotid artery angioplasty and/or stent-supported angioplasty for the treatment of carotid artery stenosis will receive neurological and neuropsychological evaluations
  Interventions: Procedure: Angioplasty; Device: Stent; Other: Neurological and neuropsychological evaluations; Procedure: Angiography
- Patients having angiography (control): Patients undergoing coronary angiography for the treatment of carotid artery stenosis will receive neurological and neuropsychological evaluations
  Interventions: Procedure: Angioplasty; Device: Stent; Other: Neurological and neuropsychological evaluations; Procedure: Angiography

INTERVENTIONS:
Procedure: Angioplasty — (non-experimental) Carotid artery angioplasty and/or stent-supported angioplasty
Device: Stent — (non-experimental) Precise™ Nitinol Self-Expanding Stent (Cordis Endovascular, Johnson & Johnson), S.M.A.R.T.® Control™ Stent (Cordis Endovascular, Johnson & Johnson), Wallstent® (Boston Scientific Medi-Tech)
Other: Neurological and neuropsychological evaluations — Clinical examinations consisting of a neurological and neuropsychological evaluation
Procedure: Angiography — (non-experimental) Coronary angiography

SUMMARY:
The purpose of this study is to determine how well patients undergoing carotid artery angioplasty and/or stent-supported angioplasty for the treatment of carotid artery stenosis will perform on a battery of tests to assess brain function before and after the procedure. This study will serve as a pilot project: (a) to determine incidence of neurologic/neuropsychometric change in patients undergoing carotid artery angioplasty and/or stent-supported angioplasty, and (b) to ascertain the time it takes for these changes to resolve.

DETAILED DESCRIPTION:
We hypothesize that the incidence of subtle neuropsychometric injury will be significantly greater than the incidence of stroke comparable to what we found in patients having carotid endarterectomy. Patients will be evaluated prospectively to determine the incidence of neurological morbidity based on both the neurologic/neuropsychometric examinations

The results of this study will serve to (a) determine incidence of neurologic/neuropsychometric morbidity for patients undergoing carotid artery angioplasty and/or stenting at ColumbiaPresbyterian Medical Center, (b) ascertain the time course of these changes, (c) identify intraprocedural markers for these changes, and (d) design protocols to evaluate the efficacy of therapeutic interventions.

Cerebral injury will be determined three ways.

First, all patients will be evaluated using a battery of neuropsychometric tests before and after the procedure. Persons presenting to the hospital on the day of the procedure, referred to hereafter as "Same Day", will be evaluated on the day of the procedure, one day after and at the 1 month follow up.

Preoperative neurological and neuropsychological evaluation will be performed. The neuropsychometric tests are designed to demonstrate general neuropsychological pathology. These tests can be divided into four types: (1) an evaluation of language, (2) an evaluation of speed of mental processing, (3) an evaluation of ability to learn using a list of words, and (4) an evaluation of visual perception requiring a patient to copy a complex figure. Before the battery is administered we will assess each patient's level of pain while sitting and standing using a 10 point Visual Analog Scale and then gauge their mood with a series called the Wong/Baker Faces Rating scale.

We will also evaluate each patient's quality of life using two well-known examinations (Telephone Interview for Cognitive Status (TICS) and Centers for Disease Control and Prevention HealthRelated Quality-of-Life 14Item Measure (CDC HRQOL14)) and a series of questions investigating how well patients are able to perform activities of daily living (ADLs) and instrumental activities of daily living (IADLs). These tests will be given at two time points, once before the surgery and then one month after surgery. We will look for changes in quality of life that may correlate with neuropsychometric test performance.

Serum levels of neuron specific enolase (NSE) and protein S100B, a neuronal enzyme and glial cell component respectively, markers of cell injury will demonstrate cerebral injury. Serum levels of TNFá (Tumor Necrosis Factor Alpha) and IL8 (Interleukin 8) will be used to evaluate the presence and degree of systemic inflammatory response.

DNA genotyping will be performed either by isolating leukocytes from blood and/or by obtaining a buccal swab sample. Normally blood is sampled via the femoral arterial catheter for assessment of hematocrit, and blood gas analysis.

Patients will undergo an intraprocedural transcranial Doppler ultrasonograph (TCD). TCD monitoring probes will be placed on the patient's head with a standard head frame after sedation, one probe on each side to measure the cerebral blood flow (CBF) velocity and determine the presence of emboli in the middle cerebral artery (MCA) on either side of the brain (Spencer Technologies, Seattle, WA). We hypothesize that there may be a relationship between emboli and subtle cognitive decline as ascertained by the battery of neuropsychometric exams. An electroencephalogram (EEG) will be applied to monitor for significant hemispheric cerebral ischemia which may occur when the balloon is inflated and occludes the artery. We routinely use EEG monitoring during carotid endarterectomy and its use exposes the patient to no risk.

ELIGIBILITY:
Inclusion Criteria:

* ability to speak English or Spanish
* scheduled to undergo carotid artery angioplasty and/or stent-supported angioplasty or coronary angiography

Exclusion Criteria:

* history of permanent neurological impairment
* Axis I psychiatric diagnosis or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Columbia University/NY Presbyterian Hospital
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2003-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Neuropsychometric Changes | Baseline to 1 day post-op
  Battery of neuropsychometric tests will assess performance pre-operatively and compare the post-operative performance at 1 day.

SECONDARY OUTCOMES:
Neuropsychometric Changes | Baseline to 1 month
  Battery of neuropsychometric tests will assess performance pre-operatively and compare the post-operative performance at 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Heyer, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, Department of Anesthesiology, New York, New York, United States

REFERENCES:
- [Background] Roubin GS, New G, Iyer SS, Vitek JJ, Al-Mubarak N, Liu MW, Yadav J, Gomez C, Kuntz RE. Immediate and late clinical outcomes of carotid artery stenting in patients with symptomatic and asymptomatic carotid artery stenosis: a 5-year prospective analysis. Circulation. 2001 Jan 30;103(4):532-7. doi: 10.1161/01.cir.103.4.532. PMID 11157718
- [Background] Theron JG, Payelle GG, Coskun O, Huet HF, Guimaraens L. Carotid artery stenosis: treatment with protected balloon angioplasty and stent placement. Radiology. 1996 Dec;201(3):627-36. doi: 10.1148/radiology.201.3.8939208.
- [Background] Diethrich EB, Ndiaye M, Reid DB. Stenting in the carotid artery: initial experience in 110 patients. J Endovasc Surg. 1996 Feb;3(1):42-62. doi: 10.1583/1074-6218(1996)0032.0.CO;2. PMID 8798126
- [Background] Wholey MH, Wholey MH, Jarmolowski CR, Eles G, Levy D, Buecthel J. Endovascular stents for carotid artery occlusive disease. J Endovasc Surg. 1997 Nov;4(4):326-38. doi: 10.1177/152660289700400402. PMID 9418194
- [Background] Henry M, Amor M, Klonaris C, Henry I, Masson I, Chati Z, Leborgne E, Hugel M. Angioplasty and stenting of the extracranial carotid arteries. Tex Heart Inst J. 2000;27(2):150-8. PMID 10928503
- [Background] Heyer EJ, Sharma R, Rampersad A, Winfree CJ, Mack WJ, Solomon RA, Todd GJ, McCormick PC, McMurtry JG, Quest DO, Stern Y, Lazar RM, Connolly ES. A controlled prospective study of neuropsychological dysfunction following carotid endarterectomy. Arch Neurol. 2002 Feb;59(2):217-22. doi: 10.1001/archneur.59.2.217. PMID 11843692
- [Background] Meyers, Philip M, Lavine, Sean D, Higashida, Randall T, Endovascular Revascularization of Carotid Artery Disease in Controversies in neurological Surgery: Neurovascular Diseases, In Press 2003.